CLINICAL TRIAL: NCT03698435
Title: (Val)Ganciclovir Therapeutic Drug Monitoring in Transplant Recipients
Brief Title: (Val)Ganciclovir TDM in Transplant Recipients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Jan-Willem C Alffenaar, Principal Investigator, Clinical pharmacologist, University Medical Center Groningen
Other Study IDs: 201800021
Record Dates: First submitted 2018-02-07; First posted 2018-10-09 (Actual); Last update posted 2019-10-10 (Actual); Status verified 2019-10

CONDITIONS: Cytomegalovirus Infections
Keywords: ganciclovir; valganciclovir; therapeutic drug monitoring; pharmacokinetics
MeSH Terms: conditions — Cytomegalovirus Infections; Multiple Acyl Coenzyme A Dehydrogenase Deficiency | interventions — Ganciclovir; Valganciclovir

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Prophylaxis: Patients who receive (val)ganciclovir for prophylaxis of cytomegalovirus
  Interventions: Drug: Ganciclovir; Drug: Valganciclovir
- Treatment: Patients who receive (val)ganciclovir for treatment of cytomegalovirus
  Interventions: Drug: Ganciclovir; Drug: Valganciclovir

INTERVENTIONS:
Drug: Ganciclovir — Intravenous ganciclovir + TDM
  Other Names: Cymevene
Drug: Valganciclovir — Oral valganciclovir + TDM
  Other Names: Valcyte

SUMMARY:
The aim of this study is to gain more insight into therapeutic drug monitoring and thus the pharmacodynamics and pharmacokinetics of ganciclovir, in the context of prophylaxis and treatment of CMV infections, in order to provide the patient with an adequate dose.

DETAILED DESCRIPTION:
Patients undergoing solid organ or stem cell transplantation are at risk of developing cytomegalovirus (CMV) infection or reactivation. The risk of CMV infection / reactivation and its severity depends on the CMV serostatus of donor and recipient. Valganciclovir (oral pro-drug of ganciclovir) prophylaxis is used to postpone CMV infection or reactivation to a later point in the post-transplantation.

CMV infection/reactivation does not always lead to clinical disease. Valganciclovir (oral) can be used when CMV DNA is detected in the blood, but patient has no or few complaints. However, in case of severe symptoms such as colitis, nephritis, hepatitis, pneumonitis, uveitis or encephalitis (active CMV disease) then ganciclovir is indicated intravenously. In clinical recovery treatment is often completed with valganciclovir.

It is important that the ganciclovir level is adequate, because too high level can lead to side effects such as cytopenia and a too low level can lead to treatment failure and resistance development. There are different dosing schedules mentioned in different sources. These schemes are based on dated literature.

The aim of (val)ganciclovir therapeutic drug monitoring (TDM) is to gain more insight into the pharmacodynamics and pharmacokinetics of ganciclovir, in the context of prophylaxis and treatment of CMV infections, in order to provide the patient with an adequate dose.

ELIGIBILITY:
Inclusion Criteria:

* Must receive ganciclovir intravenously or valganciclovir orally as routine care
* Must have received a solid organ or stem cell transplant
* Must be be 18 years or older

Exclusion Criteria:

There are no exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing solid organ or stem cell transplantation are at risk of developing cytomegalovirus (CMV) infection or reactivation. Valganciclovir (oral pro-drug of ganciclovir) prophylaxis is used to postpone CMV infection or reactivation to a later point in the post-transplantation.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-05-25 (Actual); Primary Completion 2019-11-30 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Failure of CMV treatment (with valganciclovir and ganciclovir) using viral load measurements and determining mutations in CMV kinase gene UL97 and DNA polymerase gene UL54 | 12 months after transplantation
  How many days to the development of failure of treatment? Failure of treatment is defined by increased viral load (measured in serum, whole blood, plasma in copies per mL and/or viral resistance (change of ganciclovir treatment to foscarnet treatment as a consequence, resistance is determined by resistance testing determining CMV kinase gene UL97 and DNA polymerase gene UL54 for mutations) or death due to CMV.

SECONDARY OUTCOMES:
Breakthrough CMV infection during CMV prophylaxis with valganciclovir | 12 months after transplantation
  Breakthrough CMV infection during prophylaxis with valganciclovir, time (days) to development of breakthrough CMV infection during prophylaxis
Therapeutic window | 12 months after transplantation
  How many levels are in and out of the therapeutic window (how many low and high levels)?
Successful treatment while receiving (val)ganciclovir determined by two consequtive negative viral loads | 12 months after transplantation
  The proportion of patients from CMV treatment group who have a successful CMV treatment, successful CMV treatment is defined by viral load <100 copies/mL (measured twice in a row).
(Val)ganciclovir for treatment outcomes (1) | 12 months after transplantation
  The proportion of patients from CMV treatment group who are under-dosed
(Val)ganciclovir for treatment outcomes (2) | 12 months after transplantation
  The proportion of patients from CMV treatment group who develop resistance to ganciclovir
Factors that can influence trough concentrations of (val)ganciclovir (1) | 12 months after transplantation
  Does the type of transplanted organ (liver, lungs, kidney, heart, stem cell transplant) cause high or low (val)ganciclovir trough concentrations (mg/L)? Defined therapeutic window for prophylaxis is 1-2 mg/L and for therapy is 2-4 mg/L. Number of levels which are out of the therapeutic window for different transplants.
Factors that can influence trough concentrations of (val)ganciclovir (2) | 12 months after transplantation
  Does the underlying disease for transplantation cause high or low (val)ganciclovir trough concentrations (mg/L)? Defined therapeutic window for prophylaxis is 1-2 mg/L and for therapy is 2-4 mg/L. Number of levels which are out of the therapeutic window for different underlying diseases.
Factors that can influence trough concentrations of (val)ganciclovir (3) | 12 months after transplantation
  Does dose reduction for renal failure cause increase or decrease in (val)ganciclovir trough concentrations (mg/L)? Number of levels which are out of the therapeutic window after dose reduction.

CONTACTS AND LOCATIONS:
Overall Officials: Jan-Willem Alffenaar, PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- UMCG, Groningen, Netherlands